CLINICAL TRIAL: NCT00493805
Title: Study to Evaluate Response Rates in Chronic Hepatitis C (CHC) Patients Genotype 1 With Insulin Resistance and to Assess Prolonged Treatment Duration in Late Virological Responders
Brief Title: Study of Response in Chronic Hepatitis C (CHC) Participants Genotype 1 With Insulin Resistance and Prolonged Treatment Duration in Late Responders (P04823/MK-4031-303)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04823; EudraCT number:2006-000757-21
Record Dates: First submitted 2007-06-25; First posted 2007-06-28 (Estimated); Results first posted 2011-02-09 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic; Insulin Resistance
Keywords: homeostasis model assessment of insulin resistance
MeSH Terms: conditions — Hepatitis C, Chronic; Insulin Resistance | interventions — Ribavirin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional Study arm (with insulin resistance) (Experimental): HOMA IR (homeostasis model assessment-estimated insulin resistance) of > 2
  These participants received PEG-Intron 1.5 μg /kg subcutaneously (SC) once weekly plus weight based Rebetol 800-1400 mg by mouth (PO) administered twice daily (BID) for a variable period depending on their response to treatment.
  Interventions: Drug: Combination of pegylated interferon alfa-2b and ribavirin
- Non interventional study arm (without insulin resistance) (Experimental): HOMA IR <= 2
  These participants received PEG-Intron 1.5 μg /kg subcutaneously (SC) once weekly plus weight based Rebetol 800-1400 mg PO administered twice daily (BID) for 48 weeks. (Participants are treated according to
  European labeling).
  Interventions: Drug: Combination of pegylated interferon alfa-2b and ribavirin

INTERVENTIONS:
Drug: Combination of pegylated interferon alfa-2b and ribavirin — 1. Powder for injection in Redipen (50, 80, 100, 120, and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for 12 weeks, then up to 4 weeks until HCV PCR results are available, and then for another 36 weeks(Group A) or 60 weeks (Group B) postrandomization.
  2. 200 mg capsules, oral, weight based dose of 800-1400 mg, daily for up to 12 weeks, then up to 4 weeks until HCV PCR results are available, and then for another 36 weeks (Group A) or 60 weeks (Group B) postrandomization
  Other Names: (a) SCH 54031, PEG-Intron; (b) SCH 18908, Rebetol
  Arms: Interventional Study arm (with insulin resistance)
Drug: Combination of pegylated interferon alfa-2b and ribavirin — 1. Powder for injection in Redipen (50, 80, 100, 120, and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for 48 weeks
  2. 200 mg capsules, oral, weight based dose of 800-1400 mg, daily for 48 weeks
  Other Names: (a) SCH 54031, PEG-Intron; (b) SCH 18908, Rebetol
  Arms: Non interventional study arm (without insulin resistance)

SUMMARY:
This is a Phase 3b/4, prospective, open-label, randomized, multicenter study of peginterferon alfa-2b plus ribavirin in participants with chronic hepatitis C, genotype 1. The study consists of two parts: (1) a noninterventional arm (HOMA IR <= 2) and (2) an interventional arm (HOMA IR > 2), where HOMA IR is the insulin resistance index for the participants calculated by fasting insulin (uU/mL) x [fasting glucose (mmol/L)/22.5]. Participants in the noninterventional arm are treated according to the European labeling and response rates are evaluated at Month 1 (optional), 3, 6, 12, and follow up. Participants in the interventional arm are treated with PEG-Intron 1.5 ug/kg (subcutaneous) once weekly plus weight-based REBETOL 800-1400 mg (oral capsules) daily for a variable period depending on their response at Week 12: (1) HCV-RNA positive with < 2-log drop in viral load, treatment will be discontinued; (2) HCV-RNA positive with >= 2-log drop in viral load; participants will be randomized (1:1) to Group A (stop treatment at Week 48) or Group B (stop treatment at Week 72); and (3) HCV-RNA negative, treatment will be changed to be according to the European labeling and response rates will be evaluated at Month 6, 12, and follow up. All participants will go on with their treatment after Week 12 until the results of the HCV polymerase chain reaction (PCR) are available (maximum of 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* male and female participants with newly diagnosed chronic hepatitis C
* age 18-65
* HCV-RNA positive in serum as measured by PCR
* Genotype 1
* ALT levels according to European labeling
* in women of child-bearing age, pregnancy must be excluded prior to entry into the study, and the use of a safe contraceptive device must be documented; sexually active male participants must practice a method of contraception considered acceptable (vasectomy, condom plus spermicide, plus relationship with a female partner who practices an acceptable method of contraception)
* Lab parameters:

  * Hb: >=12 g/dL (women) or >= 13 g/dL (men)
  * leukocytes >= 3,000/µL
  * thrombocytes >= 100,000/µL
  * PT/PTT/coagulation must be within normal limits or clinically acceptable to the investigator/sponsor
  * Albumin must be within normal limits or clinically acceptable to the investigator/sponsor
  * creatinine must be within normal limits or clinically acceptable to the investigator/sponsor
  * uric acid must be within normal limits or clinically acceptable to the investigator/sponsor
* antinuclear antibodies <= 1:160
* signed informed consent

Exclusion Criteria:

* refusal by women of child-bearing age or by sexually active participants to use a safe contraceptive
* breast-feeding women
* cirrhosis stage B and C according to Child-Pugh
* signs of decompensated liver disease
* confirmed co-infection with HIV or HBV
* existing psychiatric comorbidity
* alcohol abuse
* active malignant disease or suspicion or history of malignant disease within 5 previous years (except for adequately treated basal cell carcinoma)
* existing psoriasis or other dermatological disorder
* treatment with a study drug within the last 30 days
* any uncontrolled underlying medical conditions
* clinically significant ECG abnormalities and/or significant cardiovascular dysfunction within the last 6 months. In case of other suspected heart disease, a cardiological examination is required.
* any liver disorder of other genesis than the study indication (with regard to elevated iron levels, only participants with manifest hemochromatosis are excluded)
* autoimmune disorder (except LKM-positive participants).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Non Interventional Arm HOMA IR <= 2: Participants in the non-interventional arm received PegIntron at a dose of 1.5 µg /kg based on the subject's body weight at baseline visit; administrated once weekly, subcutaneously (SC) for 48 weeks together with Rebetol at a dose of 800-1400 mg based on the subject's body weight at baseline visit; administered twice daily (BID), by mouth (PO) for 48 weeks (according to European labeling). Followed by a 24-week follow up period after end of treatment.
- Interventional Arm HOMA IR > 2: Participants in the interventional arm received PegIntron at a dose of 1.5 µg /kg based on the subject's body weight at baseline visit; administrated once weekly, subcutaneously (SC) together with Rebetol at a dose of 800-1400 mg based on the subject's body weight at baseline visit; administered twice daily (BID), by mouth (PO) for 12-16 weeks until their HCV polymerase chain reaction (PCR) results are available at Week 12. At Week 12, participants with >=2 log decrease of HCV RNA were randomized to continue either for another 36 weeks (Group A- a total of 48 weeks therapy) OR for another 60 weeks (Group B- a total of 72 weeks of therapy) with a 24-week follow up. Randomization was done between Day 1 Week 17 and Day 1 Week 25.
Period: Overall Study
Arm/Group | Non Interventional Arm HOMA IR <= 2 | Interventional Arm HOMA IR > 2
Started | 17 | 42
Completed | 17 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total for Interventional Arm and Non Interventional Arm
Number analyzed (Participants) | 59
Age, Customized [Number; unit: Participants]
  Between 18 and 65 years | 59
Sex/Gender, Customized [Number; unit: Participants]
  Male | 35
  Female | 24

OUTCOME MEASURES:

1. Primary Outcome: Early Virological Response in Participants With and Without Insulin Resistance
Description: Early Virological Response (EVR) defined as HCV PCR at Week 12 either negative or at least 2 log units less than baseline in participants with and without insulin resistance.
Time Frame: At Week 12 (after start of therapy)
Population: Interventional arm: At baseline, PCR measurements for 38 out of 42 participants were available.
  Non Interventional arm: At baseline, PCR measurements for 15 out of 17 participants were available.
Measure: Number; unit: Participants
Arm/Group | Non Interventional Arm HOMA IR <= 2 | Interventional Arm HOMA IR > 2
Number analyzed (Participants) | 15 | 38
Participants | 10 | 24

2. Secondary Outcome: Sustained Virological Response (PCR 24 Weeks After End of Treatment)
Description: Sustained virological response (SVR) was defined as undetectable HCV RNA in serum at the end of follow-up (24 weeks after end of therapy) according to a polymerase chain reaction (PCR) assay.
Time Frame: Up to 24 weeks following 48 or 72 weeks of therapy
Population: Information on PCR was available for 7 participants in the non interventional study arm and 11 participants in the interventional study arm.
Measure: Number; unit: Participants
Arm/Group | Non Interventional Arm HOMA IR <= 2 | Interventional Arm HOMA IR > 2
Number analyzed (Participants) | 7 | 11
Participants | 1 | 3

ADVERSE EVENTS:
Arm/Group | Non Interventional Arm HOMA IR <=2 | Interventional Arm HOMA IR >2
Serious Adverse Events (participants affected / at risk) | 3/17 | 4/42
Other Adverse Events (participants affected / at risk) | 15/17 | 37/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Interventional Arm HOMA IR <=2 (N=17) | Interventional Arm HOMA IR >2 (N=42)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Interventional Arm HOMA IR <=2 (N=17) | Interventional Arm HOMA IR >2 (N=42)
ANAEMIA (Blood and lymphatic system disorders) | 1 (4) | 10 (28)
HAEMOGLOBINAEMIA (Blood and lymphatic system disorders) | 0 (0) | 3 (9)
LEUKOPENIA (Blood and lymphatic system disorders) | 8 (14) | 13 (34)
NEUTROPENIA (Blood and lymphatic system disorders) | 6 (13) | 12 (26)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (10)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 3 (3)
VISUAL ACUITY REDUCED (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 5 (6)
CHAPPED LIPS (Gastrointestinal disorders) | 0 (0) | 3 (4)
CHEILITIS (Gastrointestinal disorders) | 0 (0) | 5 (5)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 3 (3)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (4) | 8 (8)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 5 (5)
CHEST PAIN (General disorders) | 2 (2) | 1 (1)
FATIGUE (General disorders) | 2 (2) | 8 (8)
FEELING COLD (General disorders) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 5 (5) | 13 (14)
PAIN (General disorders) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 3 (3) | 7 (12)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 3 (3) | 14 (15)
HYPOTONIA (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 4 (6) | 5 (5)
DYSTHYMIC DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 3 (3) | 6 (7)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 (6) | 6 (6)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
NEURODERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (5) | 11 (12)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
POOR PERIPHERAL CIRCULATION (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No